CLINICAL TRIAL: NCT01061814
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate the Relative Bioavailability, Pharmacokinetics, Safety, and Tolerability of Daily, Thrice Weekly, and Weekly Dosing Regimens of Mipomersen Administered Subcutaneously to Healthy Volunteers
Brief Title: A Study to Evaluate 3 Different Dosing Regimens of Mipomersen Administered Via Subcutaneous Injections to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIPO3200309
Record Dates: First submitted 2010-01-08; First posted 2010-02-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteer
Keywords: ApoB (Apolipoprotein B); LDL (low density lipoprotein); mipomersen; ISIS301012; antisense
MeSH Terms: interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mipomersen (Experimental): 30 mg (cohort A), 70mg (cohort B) or 200mg (cohort C) SC daily
  Interventions: Drug: mipomersen
- Placebo (Placebo Comparator): 30 mg (cohort A), 70mg (cohort B), or 200mg (cohort C) SC daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mipomersen — 30 mg (cohort A), 70mg (cohort B) or 200mg (cohort C) subcutaneous (SC) dose of study drug daily for 3 weeks
  Other Names: ISIS 301012
  Arms: mipomersen
Drug: Placebo — 30 mg (cohort A), 70mg (cohort B), or 200mg (cohort C) subcutaneous (SC) dose of study drug daily for 3 weeks
  Arms: Placebo

SUMMARY:
Hypercholesterolemia is characterized by markedly elevated low density lipoproteins (LDL). Elevated LDL is a major risk factor for coronary heart disease (CHD). Mipomersen is an antisense drug that reduces a protein in the liver cells called apolipoprotein B-100 (apoB-100). ApoB-100 plays a role in producing low density lipoprotein cholesterol (LDL-C) (the 'bad' cholesterol) and moving it from the liver to one's bloodstream. High LDL-C is an independent risk factor for the development of coronary heart disease (CHD) or other diseases of blood vessels. It has been shown that lowering LDL-C reduces the risk of heart attacks and other major adverse cardiovascular events.

Mipomersen is an investigational product being studied to determine if it is safe and effective in lowering LDL-C in specific populations of patients with hypercholesterolemia.

This phase 1 study is being conducted to evaluate 3 different dosing regimens (daily, 3 times per week, or weekly) in healthy volunteers for a total of 3 weeks of dosing. Study procedures will include blood testing and physical examinations to assess the safety and tolerability of the different regimens. Tests will also be done to determine how much of the drug is present in the circulation (blood flow in the body). Specific pharmacokinetic (PK) tests on the blood samples will determine what the body does to the investigational product after it is injected, including how it is absorbed, distributed, the rate at which drug action begins and the duration of the effect.

Eligible subjects will receive study injections of either mipomersen or placebo over a 3 week period followed by a 12 week safety follow-up period.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind placebo-controlled, parallel-group, single center Phase 1 study to investigate the relative bioavailability, PK, safety, and tolerability of different sc dosing regimens of mipomersen in healthy volunteers. The bioavailability of 2 test regimens (Cohorts A and B) will be assessed relative to that of the reference treatment regimen (Cohort C). Approximately 84 subjects will be randomized equally to 1 of the 3 treatment regimens and then further randomized in a 3:1 ratio to mipomersen vs. placebo:

Cohort A/Test Treatment Regimen 1: up to 28 subjects will receive a 30 mg sc dose of study drug or matching volume of placebo daily for 3 weeks (21 doses; 630 mg total) Cohort B/Test Treatment Regimen 2: up to 28 subjects will receive a 70 mg sc dose of study drug or matching volume of placebo 3 times a week for 3 weeks (9 doses; 630 mg total) Cohort C/Reference Treatment Regimen: up to 28 subjects will receive a 200 mg sc dose of study drug or matching volume of placebo once a week for 3 weeks (3 doses; 600 mg total) Each subject will participate in a ≤ 6-week screening period, a 3-week treatment period, and a 12-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75, inclusive
* On acceptable birth control and/or partner compliant with acceptable contraceptive for 4 weeks prior to, during, and 12 weeks after the last study drug dose.
* In good overall health
* Body weight > 50 kg and body mass index (BMI) < 32 kg/m2
* Skin Type I-III based on Fitzpatrick scale

Exclusion Criteria:

* Clinically significant (CS) abnormalities in medical history, physical examination or laboratory assessments
* Positive test for human immunodeficiency virus (HIV), hepatitis B or C.
* Malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for > 1 year)
* History of rash, impetigo, or drug allergies
* Alcohol and/or drug abuse
* Receiving prescription medications within 30 days, with the exception of contraceptives; Vaccinations are not allowed beginning 3 weeks prior to the first dose of study drug until completion of the Day 28 visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs and SAEs | Assessed at each study visit through 21 weeks
Maximum plasma concentration (Cmax) | variable up to 105 days
time to maximal concentration (Tmax) | variable up to 105 days
area under the curve (AUC) based on PK profiles following the first and last dose | variable up to 105 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Anapharm, Inc., Montreal, Quebec, Canada

REFERENCES:
- [Derived] Flaim JD, Grundy JS, Baker BF, McGowan MP, Kastelein JJ. Changes in mipomersen dosing regimen provide similar exposure with improved tolerability in randomized placebo-controlled study of healthy volunteers. J Am Heart Assoc. 2014 Mar 13;3(2):e000560. doi: 10.1161/JAHA.113.000560. PMID 24627419